CLINICAL TRIAL: NCT05858788
Title: A Phase 1, Open Label, 3-treatment Period, 1-sequence, Cross-over Study to Evaluate Pharmacokinetics, Safety, and Tolerability After Single Ascending Oral Doses of SAR441566 in Healthy Adult Japanese Male Participants.
Brief Title: A Single Ascending Dose Study to Characterize the Pharmacokinetics, Safety, and Tolerability of SAR441566 in Healthy Adult Japanese Male Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PKM17860; U1111-1287-6944 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAR441566 (Experimental): Participants will receive single ascending doses of SAR441566 on day 1 of each 8-12-day cycle
  Interventions: Drug: SAR441566

INTERVENTIONS:
Drug: SAR441566 — Tablet

SUMMARY:
This is a cross-over, Phase 1, 3-treatment period single sequence study. The purpose of this study is to characterize pharmacokinetics (PK), safety, and tolerability of single ascending oral doses of SAR441566 in healthy male Japanese participants, 18-55 years of age.

DETAILED DESCRIPTION:
The duration of the study for a participant will be up to approximately 65 days.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants whose Japanese ethnicity is defined according to the following criteria: born in Japan or born outside of Japan, and are descendent of 4 ethnic Japanese grandparents who were all born in Japan.
* Male participants between the ages of 18 and 55 years, inclusive
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination including 12-lead ECG, and clinical laboratory tests)
* Body weight between 50.0 and 100.0 kg, inclusive, and body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, dermatological (including phototoxic dermatitis), osteomuscular, articular, psychiatric, systemic, ocular, immune disorders or infectious disease, or signs of acute illness.
* Receipt of live (attenuated) vaccines within 3 months and/or non live vaccines (eg, COVID-19 vaccination) within 4 weeks prior to first dose on Day 1, or planned to receive these vaccines at any time throughout the study.
* History of tuberculosis and/or a positive QuantiFERON-TB Gold (QFT) test.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B core antibody (anti-HBc Ab), anti-hepatitis C virus antibody (anti-HCV Ab), anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab), SARS-CoV-2
* Any medication within 14 days before inclusion (before first study treatment administration) or within 5 times the elimination half-life or pharmacodynamic half-life of the medication whichever the longest.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Assessment of plasma pharmacokinetic (PK) parameters for SAR441566: Cmax | From Day 1 to Day 5 of each period (5 days per period)
  Maximum plasma concentration observed
Assessment of plasma pharmacokinetic (PK) parameters for SAR441566: AUClast | From Day 1 to Day 5 of each period (5 days per period)
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time Tlast (AUClast)
Assessment of plasma pharmacokinetic (PK) parameters for SAR441566: AUC | From Day 1 to Day 5 of each period (5 days per period)
  Area under the plasma concentration versus time curve extrapolated to infinity (AUC)

SECONDARY OUTCOMES:
Number of participants with adverse events (AE) and treatment-emergent adverse events (TEAEs) | Up to end of study visit (which will occur at latest day 37 of study)
  Assessment of adverse events (AE) / treatment-emergent adverse events (TEAE) including Serious AE and AE of Special Interest

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Parexel International-Site Number:8400001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- See also: PKM17860 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25330&tenant=MT_SNY_9011